CLINICAL TRIAL: NCT05318872
Title: Preliminary Evaluation of the Analytical Performance of the ENDOSWIR Medical Device (DM-DIV) Versus Anatomical Pathology Examination in Patients Operated for Squamous Cell Carcinoma of Upper Aerodigestive Tract: Prospective Pilot Study
Brief Title: Prospective Evaluation of ENDOSWIR Device Versus Pathology for Squamous Cell Carcinoma of Upper Aerodigestive Tract (ENDOSWIR-VADS)
Acronym: ENDOSWIR-VADS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institute for Advanced Biosciences (IAB), Grenoble (Unknown); Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Other Study IDs: 38RC22.0028
Record Dates: First submitted 2022-03-21; First posted 2022-04-08 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and neck neoplasms; Fluorescence; Short Wave Infra-Red
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ENT cancers: patients with ENT cancer in the active care line for who a surgical resection is planned.
  Interventions: Device: ENDOSWIR

INTERVENTIONS:
Device: ENDOSWIR — Patients were enrolled for surgery of their cancer and give their consents to the participation to that study. Characteristics of anonymized patient (sex, age, medical history, and tumoral characteristics) will be collected. During surgery, the excisional specimen will be sent in a fresh state for pathological examination (gold standard). The pathologist will determine 10 zones on a cross-section of the specimen which will be analyzed by SWIR, and compared between the two techniques.

SUMMARY:
A new medical optical device named ENDOSWIR is tested to determine its ability to determine if tissues are cancer or normal tissue on ex-vivo condition for specimen of ENT squamous cell cancers.

DETAILED DESCRIPTION:
In vivo short infrared imaging is a real-time, sensitive technique that can be used in the operating room during surgical removal of tumors.

It is essential in the surgery of cancers of the upper aerodigestive tract to be in healthy margins in order to avoid heavier surgical resumption or complementary treatments such as radiotherapy.

The optical imaging device in the short infrared range called ENDOSWIR and tested on tonsil samples has shown its safety on the analysis of tissues and seems to be promising for the detection of tumor tissues or, on the contrary, their absence in the resection margins (animal studies).

The principal objective is to determine the ability of the ENDOSWIR DM-DIV to distinguish healthy tissue from tumor tissue on an ENT squamous cell carcinoma specimen by Concordance rate (in %) between the ENDOSWIR result and the final pathology examination of each tissue portion of a subject (8 per subject)..

secondary objectives are : to demonstrate that analysis of a sample using the ENDOSWIR device is faster than extemporaneous analysis, the safety of SWIR. An ancillary analysis of areas of particular interest such as resection margins or carcinoma in situ/dysplasia areas etc...

ELIGIBILITY:
Inclusion Criteria:

* ENT cancer (buccal or oropharyngeal) for which a surgical resection is planned
* affiliated to the social security
* Having given his non-opposition to participate in the trial.

Exclusion Criteria:

* Patient protected by law (minor, pregnant or breastfeeding woman, patient under guardianship, subject deprived of liberty or hospitalized under restraint).
* Patients who have received radiotherapy treatment in the VADS area
* Patient with a history of VADS cancer or a synchronous location of VADS cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is selected from the subjects operated on for ENT carcinoma in a programmed manner and as part of the management at the CHUGA.
  The active file of the CHUGA for an exeresis of squamous cell carcinoma of the oral cavity or oropharynx is about 1 subject per week which should allow to finalize the project in 6 months by supposing that it will be possible to include 50% of the subjects.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-04-11 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Ability of the ENDOSWIR in-vitro diagnostic medical device to distinguish healthy tissue from tumoral tissue on an ENT squamous cell carcinoma resection | 1 day
  Concordance rate (in %) between the ENDOSWIR result and the final pathological examination.

SECONDARY OUTCOMES:
Demonstration that analysis of a sample using the ENDOSWIR device is faster than extemporaneous analysis | 1 day
  Time (in minutes) for ENDOSWIR data acquisition and processing.
Demonstration of the safety of SWIR. | 1 day
  No perceptible tissue change on the SWIR exposed sample
Ancillary analysis of special interest areas | 1 day
  Concordance rate and descriptive qualitative analysis between the ENDOSWIR result and the final pathological examination of tissue portions located in a subject's areas of special interest

CONTACTS AND LOCATIONS:
Overall Officials: Christian Righini, MD, PhD, Principal Investigator — CHU Grenoble Alpes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wilson RH, Nadeau KP, Jaworski FB, Tromberg BJ, Durkin AJ. Review of short-wave infrared spectroscopy and imaging methods for biological tissue characterization. J Biomed Opt. 2015 Mar;20(3):030901. doi: 10.1117/1.JBO.20.3.030901. PMID 25803186
- [Result] Kenry, Duan Y, Liu B. Recent Advances of Optical Imaging in the Second Near-Infrared Window. Adv Mater. 2018 Nov;30(47):e1802394. doi: 10.1002/adma.201802394. Epub 2018 Sep 4. PMID 30182451
- [Result] Hu Z, Fang C, Li B, Zhang Z, Cao C, Cai M, Su S, Sun X, Shi X, Li C, Zhou T, Zhang Y, Chi C, He P, Xia X, Chen Y, Gambhir SS, Cheng Z, Tian J. First-in-human liver-tumour surgery guided by multispectral fluorescence imaging in the visible and near-infrared-I/II windows. Nat Biomed Eng. 2020 Mar;4(3):259-271. doi: 10.1038/s41551-019-0494-0. Epub 2019 Dec 23. PMID 31873212
- [Result] Schols RM, ter Laan M, Stassen LP, Bouvy ND, Amelink A, Wieringa FP, Alic L. Differentiation between nerve and adipose tissue using wide-band (350-1,830 nm) in vivo diffuse reflectance spectroscopy. Lasers Surg Med. 2014 Sep;46(7):538-45. doi: 10.1002/lsm.22264. Epub 2014 Jun 4. PMID 24895321